CLINICAL TRIAL: NCT00781456
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy of DR-105 Compared to Placebo For the Management of Menstrually-Related Migraine Headaches.
Brief Title: A Multicenter Study to Evaluate the Efficacy of a 91-Day Extended Cycle Oral Contraceptive for Menstrually-Related Migraine Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DR-105-201
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Migraine
Keywords: Migraine headache; menstrual; oral contraceptive; Menstrually-Related Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Seasonique

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 91-day Levonorgestrel Oral Contraceptive (Experimental): Participants received 12 weeks (84 consecutive days) of active combination tablets containing 150 µg levonorgestrel (LNG)/30 µg ethinyl estradiol (EE), followed by 7 days of 10 µg EE monotherapy, for a total of 13 weeks.
  Interventions: Drug: 91-day Levonorgestrel Oral Contraceptive
- Placebo (Placebo Comparator): Participants received placebo, 12 weeks (84 consecutive days) of inactive tablets, followed by an additional 7 days of inactive tablets, for a total of 13 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 91-day Levonorgestrel Oral Contraceptive — 91-day treatment consisting of 84 blue combination tablets containing 150 µg LNG/30 µg EE and 7 yellow tablets containing 10 µg EE.
  Other Names: Seasonique; DR-105
  Arms: 91-day Levonorgestrel Oral Contraceptive
Drug: Placebo — 1 tablet daily to match experimental arm
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the efficacy of a 91-day extended cycle oral contraceptive compared to placebo for decreasing the frequency and severity of menstrually-related migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, non-pregnant, non-lactating
* History of migraine headaches without aura for at least 6 months
* History of migraine headaches associated with menstruation
* Others as directed by FDA-approved protocol

Exclusion Criteria:

* History of migraine headaches with aura or focal neurological symptoms
* Any contraindication to the use of oral contraceptives
* Others as dictated by FDA-approved protocol

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Research Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (22):
- United States (22):
  - Teva Investigational Site, La Mesa, California
  - Duramed Investigational Site, San Diego, California
  - Teva Investigational Site, San Diego, California
  - Duramed Investigational Site, San Francisco, California
  - Duramed Investigational Site, Washington D.C., District of Columbia
  - Duramed Investigational Site, West Palm Beach, Florida
  - Teva Investigational Site, Savannah, Georgia
  - Duramed Investigational Site, Edison, New Jersey
  - Duramed Investigational Site, New York, New York
  - Teva Investigational Site, Winston-Salem, North Carolina
  - Teva Investigational Site, Tulsa, Oklahoma
  - Teva Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Teva Investigational Site, Uniontown, Pennsylvania
  - Teva Investigational Site, Columbia, South Carolina
  - Teva Investigational Site, Hilton Head, South Carolina
  - Teva Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Dallas, Texas
  - Teva Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Virginia Beach, Virginia
  - Duramed Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 304 women with menstrually related migraine were screened for enrollment at 37 study centers in the United States. Of the 304 screened, 109 women at 23 centers met entry criteria and were considered eligible for enrollment into the study.
Period: Overall Study
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Started | 58 | 51
Received Study Drug | 57 | 49
Completed | 37 | 35
Not Completed | 21 | 16
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Protocol Violation | 4 | 1
Not completed — Noncompliance With Protocol | 1 | 1
Not completed — Lost to Follow-up | 10 | 5
Not completed — Other Reason, Unknown | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population includes all randomly assigned and treated participants who had at least 1 week of postbaseline migraine data.
Groups:
- Total: Total of all reporting groups
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo | Total
Number analyzed (Participants) | 54 | 45 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (4.70) | 27.4 (3.83) | 27.1 (4.32)
Gender [Count of Participants; unit: Participants]
  Female | 54 | 45 | 99
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28 | 23 | 51
  Black | 11 | 9 | 20
  Asian | 1 | 1 | 2
  Hispanic or Latino | 14 | 10 | 24
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 50% Reduction in Migraine Frequency During the Treatment Period
Description: The number of participants with at least 50% reduction in migraine frequency (average weekly number of migraine episodes) through the end of the 91-day treatment period compared with Baseline (the 25- to 35-day baseline qualification period). Participants recorded the incidence, timing and intensity of migraines in a migraine diary during the prequalification period and throughout the 91-day treatment period.
Time Frame: Baseline (25-35 days before Day 1) and Days 1-91
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 54 | 45
percentage of participants | 48.1 | 48.9
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Test type: Superiority or Other; p = 0.954, Regression, Logistic; Logistic regression model with terms of treatment, weekly baseline migraine frequency, and center included in the model; Odds Ratio, log = 0.02, 95% CI 2-sided [-0.82 to 0.87], Standard Error of Mean 0.43 — 91-day Levonogestrel Oral Contraceptive versus placebo. Treatment Difference was estimated using logistic regression for the proportion of participants with >=50% reduction in migraine frequency during the treatment period

2. Secondary Outcome: Percentage of Participants With ≥ 50% Reduction in Migraine Frequency During the First, Second and Third Months
Description: The percentage of participants with at least 50% reduction in migraine frequency (average weekly number of migraine episodes) compared to Baseline at each month of the treatment period.
Time Frame: Baseline, Month1, Month 2 and Month 3
Population: Intent-to-treat population with available data. N indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 54 | 45
percentage of participants
  First Month (N=54, 45) | 42.6 | 37.8
  Second Month (N=51, 44) | 62.7 | 52.3
  Third Month (N=40, 37) | 60.0 | 64.9
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants with a reduction of 50% or more in migraine frequency during the first month of treatment; Test type: Superiority or Other; p = 0.479, Regression, Logistic — No adjustment for multiple comparisons was performed; Logistic regression model with terms of treatment, baseline weekly migraine frequency and center included in the model; Odds Ratio, log = 0.31, 95% CI 2-sided [-0.55 to 1.17], Standard Error of Mean 0.44 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants with a reduction of 50% or more in migraine frequency during the second month of treatment; Test type: Superiority or Other; p = 0.256, Regression, Logistic — No adjustment for multiple comparisons was performed; Logistic regression model with terms of treatment, baseline weekly migraine frequency and center included in the model; Odds Ratio, log = 0.50, 95% CI 2-sided [-0.36 to 1.37], Standard Error of Mean 0.44 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants with a reduction of 50% or more in migraine frequency during the third month of treatment; Test type: Superiority or Other; p = 0.788, Regression, Logistic — No adjustment for multiple comparisons was performed; Logistic regression model with terms of treatment, baseline weekly migraine frequency and center included in the model; Odds Ratio, log = -0.14, 95% CI 2-sided [-1.16 to 0.88], Standard Error of Mean 0.52 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Average Migraine Severity
Description: Migraine severity was recorded by participants in the Baseline qualification diary and study migraine diary during the treatment period. Participants could report a severity of none (score = 0), mild (1), moderate (2), or severe (3). In general, if a headache was mild, daily activities could be resumed and little to no medication was taken. Moderate headaches required medication and effected daily activities. Severe headaches were debilitating and required medication.
  Average migraine severity is defined as the sum of the severity ratings divided by the total number of migraine episodes reported during the observation period (for example, Baseline, First Month, Second Month, Third Month, and 91-Day Treatment Period). A negative change from Baseline score indicates improvement in severity.
Time Frame: Baseline and Month 1, Month 2 and Month 3
Population: Intent-to-treat population with available data. N indicates the number of participants with available data at each time period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 54 | 45
units on a scale
  91-Day Treatment Period (N=54, 45) | -0.37 (0.097) | -0.18 (0.109)
  First Month (N=54, 45) | -0.55 (0.138) | -0.52 (0.154)
  Second Month (N= 51, 44) | -0.98 (0.158) | -0.72 (0.173)
  Third Month (N=40, 37) | -1.06 (0.190) | -0.66 (0.197)
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of change from Baseline in migraine severity during the 91-day treatment period; Test type: Superiority or Other; p = 0.182, ANCOVA; Treatment comparison was performed using an analysis of covariance model with baseline average migraine severity and center as covariates; Odds Ratio, log = -0.19, 95% CI 2-sided [-0.47 to 0.09] — 91-day Levonogestrel Oral Contraceptive versus placebo
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of change from Baseline in migraine severity during the first month of treatment; Test type: Superiority or Other; p = 0.853, ANCOVA; [statistical method as in outcome 3, analysis 1]; Odds Ratio, log = -0.04, 95% CI 2-sided [-0.71 to 0.19] — 91-day Levonogestrel Oral Contraceptive versus placebo
Statistical Analysis 3: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of change from Baseline in migraine severity during the second month of treatment; Test type: Superiority or Other; p = 0.249, ANCOVA; [statistical method as in outcome 3, analysis 1]; Odds Ratio, log = -0.26, 95% CI 2-sided [-0.71 to 0.19] — 91-day Levonogestrel Oral Contraceptive versus placebo
Statistical Analysis 4: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of change from Baseline in migraine severity during the third month of treatment; Test type: Superiority or Other; p = 0.119, ANCOVA; [statistical method as in outcome 3, analysis 1]; Odds Ratio, log = -0.40, 95% CI 2-sided [-0.90 to 0.10] — 91-day Levonogestrel Oral Contraceptive versus placebo

4. Secondary Outcome: Percentage of Participants Who Required Rescue Medications During the Study Period
Description: Participants recorded use of rescue medications for migraines in the migraine diary during the course of study treatment.
Time Frame: Baseline, Month 1, Month 2 and Month 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 54 | 45
percentage of participants
  Baseline (N=54, 45) | 85.2 | 75.6
  First Month (N=54, 45) | 63.0 | 55.6
  Second Month (N=51, 44) | 45.1 | 54.5
  Third Month (N=40, 37) | 35.0 | 62.2
  During the 91-day treatment period (N=54, 45) | 72.2 | 75.6
Statistical Analysis 1: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants requiring rescue medication during the first month of treatment; Test type: Superiority or Other; p = 0.457, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants requiring rescue medication during the second month of treatment; Test type: Superiority or Other; p = 0.361, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants requiring rescue medication during the third month of treatment; Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: 91-day Levonorgestrel Oral Contraceptive vs Placebo; Comparison of percentage of participants requiring rescue medication during the 91-day treatment period; Test type: Superiority or Other; p = 0.709, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Migraine Disability Assessment
Description: The migraine disability assessment (MIDAS) test is used to determine how severely migraines affect a patient's life. Participants were asked five questions about how often their headaches limited their ability to go to work or school, to do household work or to do family or leisure activities in the past 3 months.
  The MIDAS score equals the sum of the days answered for each question and ranges from 0 (no disability) to approximately 270 (severe disability; the upper bound is dependent on the number of days a participant would plan to work or participate in other activities).
  The MIDAS score is classified into four grades of severity:
  * 0 to 5: MIDAS Grade I, Little or no disability
  * 6 to 10: MIDAS Grade II, Mild disability
  * 11 to 20: MIDAS Grade III, Moderate disability
  * 21+: MIDAS Grade IV, Severe disability
Time Frame: Baseline and Week 15
Population: Intent-to-treat population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 46 | 40
units on a scale | -7.8 (16.26) | -8.5 (10.65)

6. Secondary Outcome: Change From Baseline in Headache Impact Test
Description: The Headache Impact Test (HIT) is a tool used to measure the impact headaches have on patients' ability to function on the job, at school, at home and in social situations.
  HIT-6 consists of 6 questions each scored on a scale from Never (6 points) to Always (13 points). The total score ranges from 36 to 78 with higher scores indicating greater impact on life.
  There was an error in administration of the HIT-6 in this study. Question 6 was not administered, and question 3 from the MIDAS was included instead. Therefore, the total score of the HIT-6 could not be calculated.
Time Frame: Baseline and Week 15
Population: Analysis was not performed due to an error in the administration of the test.
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant and which does not necessarily have to have a causal relationship with this treatment or clinical study.
  The following definitions were used to assess AE severity: Mild: Awareness of signs or symptoms, but they are easily tolerated; Moderate: Enough discomfort to cause interference with usual activity; Severe: Incapacitating, with inability to perform usual activity.
  Relationship to study drug was assessed as either: None: Causal relationship can be ruled out; Possibly: Causal relationship at least reasonably possible, i.e. relationship cannot be ruled out; Definitely: Causal relationship is certain.
  A serious adverse event (SAE) is one that met any one of the following criteria:
  * Fatal or life threatening
  * Requires or prolongs in patient hospitalization
  * Results in persistent or significant disability/incapacity
  * Congenital anomaly / birth defect
  * Important medical event.
Time Frame: Up to 15 weeks
Population: Safety population, consisting of all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 57 | 49
participants
  Any adverse event | 32 | 17
  Mild adverse event | 11 | 2
  Moderate adverse event | 17 | 10
  Severe adverse event | 4 | 5
  Adverse event not related to study drug | 11 | 6
  Adverse event possibly related to study drug | 20 | 11
  Adverse event related to study drug | 1 | 0
  Deaths | 0 | 0
  Other serious adverse event | 0 | 0
  Withdrawn due to adverse event | 3 | 3

8. Secondary Outcome: Mean Number of Days of Bleeding or Spotting
Description: Bleeding and spotting were recorded by participants in the migraine diary during the 91-day treatment period.
Time Frame: 91-day treatment period
Population: Safety population with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Number analyzed (Participants) | 56 | 47
days | 21.2 (19.58) | 15.5 (7.73)

ADVERSE EVENTS:
Time Frame: Up to 15 weeks
Arm/Group | 91-day Levonorgestrel Oral Contraceptive | Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/49
Other Adverse Events (participants affected / at risk) | 21/57 | 11/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 91-day Levonorgestrel Oral Contraceptive (N=57) | Placebo (N=49)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 11 (18) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (6) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 5 (7) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 6 (7) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.